CLINICAL TRIAL: NCT00002494
Title: HIGH INTENSITY, BRIEF DURATION CHEMOTHERAPY FOR DIFFUSE SMALL NONCLEAVED CELL LYMPHOMA AND THE L-3 SUBTYPE OF ALL: A PILOT STUDY OF A MULTIDRUG REGIMEN
Brief Title: Combination Chemotherapy in Treating Patients With Non-Hodgkin's Lymphoma or Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9251; U10CA031946 (NIH); CLB-9251; CDR0000077643 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-04-06 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Leukemia; Lymphoma
Keywords: untreated adult acute lymphoblastic leukemia; L3 adult acute lymphoblastic leukemia; stage I adult Burkitt lymphoma; stage II adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Burkitt Lymphoma | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Etoposide; Ifosfamide; Leucovorin; Mesna; Methotrexate; Prednisone; Hydrocortisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination therapy (Experimental): Patients receive combination therapy as described in the study description. All patients must complete at least the first 3 courses of chemotherapy. Courses 2 and 3 each repeat 3 times in the absence of disease progression or unacceptable toxicity. On days 134-139, patients who have had prior bone marrow involvement receive cranial radiation therapy. Patients who achieve less than a complete response and who have an HLA-matched sibling should undergo allogeneic bone marrow transplant on protocol CLB-9113. Patients are followed monthly for 6 months, every 2 months for 18 months, every 6 months for 2 years, and thereafter for survival.
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: leucovorin calcium; Drug: mesna; Drug: methotrexate; Drug: prednisone; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: leucovorin calcium
Drug: mesna
Drug: methotrexate
Drug: prednisone
Drug: therapeutic hydrocortisone
Drug: vincristine sulfate
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and alternating regimens of chemotherapy in treating patients who have non-Hodgkin's lymphoma or acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and disease free survival of HIV seronegative patients with diffuse small noncleaved cell lymphoma or L3 acute lymphocytic leukemia when treated with high intensity, brief duration combination chemotherapy: alternating courses of ifosfamide/cytarabine/etoposide and cyclophosphamide/doxorubicin, each with methotrexate/vincristine/dexamethasone. II. Determine the toxicity of these regimens in HIV negative patients.

OUTLINE: Patients are stratified by participating institution and disease type (diffuse small noncleaved cell lymphoma vs L3 ALL). Patients receive cyclophosphamide IV over 5-10 minutes on days 1 through 5 and oral prednisone on days 1 through 7, followed by alternating courses of: 2) ifosfamide IV over 1 hour on days 8 through 12, methotrexate IV over 24 hours on day 8; leucovorin calcium IV over 36 hours after initiation of methotrexate, then IV (or orally as tolerated, after the first 24 hours) every 6 hours until the serum methotrexate level is below 5 x 10 to the minus eighth M; vincristine IV on day 8; cytarabine IV over 48 hours and etoposide IV over 60 minutes on days 11 and 12; and oral dexamethasone on days 8 through 12, plus triple intrathecal therapy (TIT) with methotrexate, cytarabine, and hydrocortisone on days 8 and 12, and 3) cyclophosphamide IV over 5-10 minutes on days 29 through 33; methotrexate IV over 24 hours and vincristine IV on day 29; leucovorin calcium IV over 36 hours after initiation of methotrexate, then IV (or orally as tolerated, after the first 24 hours) every 6 hours until the serum methotrexate level is below 5 x 10 to the minus eighth M; doxorubicin IV on days 32 and 33; and oral dexamethasone on days 29 through 33, plus TIT on day 29, with doses as above. Patients with CNS disease at diagnosis continue TIT once weekly until the CSF clears, then weekly for 4 more weeks. TIT must be completed prior to initiation of radiotherapy. All patients must complete at least the first 3 courses of chemotherapy. Courses 2 and 3 each repeat 3 times in the absence of disease progression or unacceptable toxicity. On days 134-139, patients who have had prior bone marrow involvement receive cranial radiation therapy. Patients who achieve less than a complete response and who have an HLA-matched sibling should undergo allogeneic bone marrow transplant on protocol CLB-9113. Patients are followed monthly for 6 months, every 2 months for 18 months, every 6 months for 2 years, and thereafter for survival.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically documented diffuse small noncleaved cell lymphoma (category J by IWF) of any stage Nodal or abdominal masses with less than 25% lymphoblasts in marrow are defined as lymphoma OR Histologically documented L3 acute lymphocytic leukemia (ALL) Greater than 25% lymphoblasts in marrow is defined as ALL, regardless of presence of bulky nodal disease Lymphoma requirements include: Documentation of lymphadenopathy, splenomegaly, or hepatomegaly, presence or absence of abdominal masses, and presence or absence of B symptoms Measurable disease other than ascites and pleural effusions, bony disease, and CNS lesions Bidimensionally measurable mass on physical exam, x-ray, or CT, or MRI OR Clearly defined hepatic mass greater than 3.5 cm on CT, MRI, or ultrasound considered to represent lymphoma OR Histologically documented hepatic lymphoma with the liver extending more than 5 cm below the costal margin on quiet respiration ALL requirements include: Documentation of monoclonal surface immunoglobulin by surface immunophenotyping Lymph node biopsy strongly recommended for patients with obvious marrow involvement Disease labeled L3 but also manifested by lymphadenopathy must be evaluated as is lymphoma (see above)

PATIENT CHARACTERISTICS: Age: 15 and over Performance status: Any status Life expectancy: At least 2 years Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 times normal (unless further elevation is directly attributable to malignancy) Renal: Creatinine no greater than 1.5 times normal (unless further elevation is directly attributable to malignancy) Cardiovascular: No uncontrolled or severe cardiovascular disease, e.g.: No myocardial infarction within the past 6 months No congestive heart failure Other: HIV negative No active, uncontrolled bacterial, viral, or fungal infection No active, uncontrolled duodenal ulcer No other serious medical illness No serious psychiatric condition that would preclude informed consent or protocol compliance No second malignancy within 5 years except: Curatively treated carcinoma in situ of the cervix Curatively treated basal cell carcinoma Not pregnant Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY: Biologic: No concurrent growth factors Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: No concurrent palliative radiotherapy Surgery: Not specified Other: No prior therapy

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 1992-05; Primary Completion 2004-03 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
complete response | up to 5 years post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lee, MD, Study Chair — Central Maryland Oncology Center
Locations (23):
- United States (23):
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Rizzieri DA, Johnson JL, Niedzwiecki D, Lee EJ, Vardiman JW, Powell BL, Barcos M, Bloomfield CD, Schiffer CA, Peterson BA, Canellos GP, Larson RA. Intensive chemotherapy with and without cranial radiation for Burkitt leukemia and lymphoma: final results of Cancer and Leukemia Group B Study 9251. Cancer. 2004 Apr 1;100(7):1438-48. doi: 10.1002/cncr.20143. PMID 15042678
- [Result] Lee EJ, Petroni GR, Schiffer CA, Freter CE, Johnson JL, Barcos M, Frizzera G, Bloomfield CD, Peterson BA. Brief-duration high-intensity chemotherapy for patients with small noncleaved-cell lymphoma or FAB L3 acute lymphocytic leukemia: results of cancer and leukemia group B study 9251. J Clin Oncol. 2001 Oct 15;19(20):4014-22. doi: 10.1200/JCO.2001.19.20.4014. PMID 11600602